CLINICAL TRIAL: NCT00003046
Title: Phase I Study of Intraperitoneal Recombinant Human Interleukin-12 (rhIL-12) in Patients With Peritoneal Carcinomatosis, Associated With Mullerian and Gastrointestinal Carcinomas
Brief Title: Interleukin-12 in Treating Patients With Cancer in the Abdomen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID97-027; P30CA016672 (NIH); MDA-ID-97027 (Other: UT MD Anderson Cancer Center); NCI-T97-0034; CDR0000065681 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-02-19 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Anal Cancer; Colorectal Cancer; Gallbladder Cancer; Gastric Cancer; Pancreatic Cancer
Keywords: anal cancer; carcinoma of the appendix; colorectal cancer; extrahepatic bile duct cancer; gallbladder cancer; gastric cancer; gastrointestinal carcinoid tumor; malignant mesothelioma; pancreatic cancer; small intestine cancer; stage IV colon cancer; stage IV gastric cancer; recurrent gastric cancer; recurrent pancreatic cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage IV anal cancer; recurrent anal cancer; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; advanced malignant mesothelioma; recurrent malignant mesothelioma; small intestine adenocarcinoma; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Anus Neoplasms; Colorectal Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Appendiceal Neoplasms; Bile Duct Neoplasms; Mesothelioma, Malignant; Colonic Neoplasms; Rectal Neoplasms | interventions — Interleukin-12 Subunit p35

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interleukin-12 (Experimental)
  Interventions: Biological: Recombinant Interleukin-12

INTERVENTIONS:
Biological: Recombinant Interleukin-12 — Intraperitoneal over 30 minutes once weekly for 4 weeks, repeats every 4 weeks for up to 6 courses
  Other Names: Intraperitoneal Recombinant Human Interleukin-12; rhIL-12

SUMMARY:
RATIONALE: Interleukin-12 may kill tumor cells by stimulating a person's white blood cells to kill cancer cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-12 in treating patients with cancer in the abdomen.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of intraperitoneal interleukin-12 in patients with Mullerian carcinoma (closed to accrual as of 8/23/01), gastrointestinal carcinoma, or peritoneal mesothelioma (closed to accrual as of 8/23/01). II. Determine the qualitative and quantitative toxicity and reversibility of toxicity of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients receive intraperitoneal interleukin-12 over 30 minutes once weekly for 4 weeks. Treatment repeats every 4 weeks for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients with stable or responsive disease may receive an additional 6 courses. Patients receive escalating doses of intraperitoneal interleukin-12 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is established, additional patients are accrued to receive interleukin-12 at the recommended dose.

PROJECTED ACCRUAL: Approximately 20-40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed Mullerian carcinoma (ovarian epithelial or peritoneal carcinoma) (closed to accrual as of 8/23/01) OR Gastrointestinal cancer with abdominal carcinomatosis OR Peritoneal mesothelioma (closed to accrual as of 8/23/01) Must have received an adequate course of any platinum-based chemotherapy regimen for ovarian cancer with evidence of intraabdominal disease Must have received an adequate course of fluorouracil-based treatment for metastatic colon cancer Intact primary gastrointestinal tumor allowed if not at risk of obstruction and/or bleeding Abdominal lesions must be less than 10 cm Extraperitoneal lesions must be less than 2 cm No hepatic disease No clinically significant pleural effusion (controlled by pleurodesis allowed) No brain metastases No significant adhesions or symptoms of obstruction

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL (transfusion allowed) Lymphocyte count at least 800/mm3 Hepatic: See Disease Characteristics Bilirubin no greater than 1.5 mg/dL SGOT or SGPT less than 2.5 times upper limit of normal Albumin at least 3.5 g/dL Hepatitis B and C negative Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No significant heart disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Loss of no more than 10% of body weight over a 4 month period No overt autoimmune disease No active ulcer disease No prior inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)

PRIOR CONCURRENT THERAPY: Biologic therapy: No other concurrent immunotherapy Chemotherapy: At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered No concurrent chemotherapy Endocrine therapy: No chronic steroid therapy Radiotherapy: At least 3 months since prior localized radiotherapy (e.g., pelvic or small field) and recovered No radiotherapy to whole abdomen No concurrent radiotherapy Surgery: Recovered from prior surgery At least 3 weeks since prior major abdominal surgery At least 2 weeks since prior laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 1997-08; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Intraperitoneal Interleukin-12 | 4 weeks
  MTD found in absence of unacceptable toxicity or disease progression with each 4 week treatment cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Lenzi, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Lenzi R, Kudelka AP, Veschraegen C, et al.: Intraperitoneal (IP) bioimmunologic responses in patients with ovarian and gastrointestinal cancers at a low toxicity dosing schedule of IP recombinant interleukin-12 (rhIL-12). [Abstract] Proc Am Assoc Cancer Res 40: A3778, 573, 1999.
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org